CLINICAL TRIAL: NCT01024517
Title: An Open Label Study to Compare the Oral Bioavailability of a Solid Dose Formulation of GLPG0259 Relative to an Oral Solution After Single-dose Intake in Healthy Subjects and to Evaluate the Effect of Food on the Solid Dose Formulation.
Brief Title: GLPG0259 Solid Formulation Bioavailability and Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos NV
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GLPG0259-CL-103
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single oral dose, solution (Experimental)
  Interventions: Drug: GLPG0259 solution
- Single oral dose, solid, fasted (Experimental)
  Interventions: Drug: GLPG0259
- Single oral dose, solid, fed. (Experimental)
  Interventions: Drug: GLPG0259

INTERVENTIONS:
Drug: GLPG0259 solution — single oral dose, GLPG0259, 50 mg oral solution
  Arms: Single oral dose, solution
Drug: GLPG0259 — single oral dose, GLPG0259, 50 mg solid formulation
  Arms: Single oral dose, solid, fasted; Single oral dose, solid, fed.

SUMMARY:
The purpose of the study is to compare the pharmacokinetics of GLPG0259 as a solid dosage formulation (with and without food)and an oral solution, and to assess its safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Bioavailability of a solid dosage formulation of GLPG0259 (with/without food) compared to an oral solution of GLPG0259. | up to 96 hours postdose

SECONDARY OUTCOMES:
Safety and tolerability of GLPG0259 | up to 96 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Johan Beetens, PharmD, PhD, Study Director — Galapagos NV; Wouter Haazen, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium